CLINICAL TRIAL: NCT02102009
Title: Impact of Nutritional Support With an Complete Formula on Nutritional Status and Respiratory Function in Adult Patients Malnourished or at Risk of Malnutrition and Chronic Respiratory Disease..
Brief Title: Nutritional Supplementation in Adults With Chronic Respiratory Disease
Acronym: OFOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Ordesa (Industry)
Collaborators: Peruvian Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OFOS-01-012
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Malnutrition; Pulmonary Disease, Chronic Obstructive; Other Pulmonary Disease, Chronic Obstructive
Keywords: Malnutrition; Dietary supplement; Nutritional supplement; Complete enteral formula; COPD
MeSH Terms: conditions — Malnutrition; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitafos (Experimental): Complete enteral formula
  Interventions: Dietary Supplement: Complete enteral formula
- Dietary Advise (Active Comparator): Dietary advise according to the hospital routine clinical practice.
  Interventions: Other: Dietary Advise

INTERVENTIONS:
Dietary Supplement: Complete enteral formula — Product: Complete nutritional formula in powder enriched with key nutrients to be administered orally (200 ml of water per 57 g product).
  Time of intervention: 3 months.
  Other Names: Vitafos; Vitafos Adultos; Vitafos Vainilla
  Arms: Vitafos
Other: Dietary Advise — Patients will receive the usual dietary advise in these patients according hospital clinical practice .
  Arms: Dietary Advise

SUMMARY:
The purpose of this study is to determine whether nutritional support with a complete formula is effective to improve malnutrition and respiratory function in patients with chronic pulmonary disease compared to the standard hospital dietary advise.

DETAILED DESCRIPTION:
This is a unicenter, controlled, randomized, prospective, parallel-group, open-label study to evaluate the effect of a nutritional formula on nutritional status, pulmonary function and quality of life. Adult patients will be randomized to receive the nutritional formula or to follow the standard hospital' dietetic recommendations during 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years.
* Patient from Clínica San Gabriel or Clínica San Pablo Surco, inpatient or outpatient.
* Patients with chronic pulmonary disease (including bronchiectasis, tuberculosis specific sequel, fibrothorax, diffuse interstitial lung disease, COPD).
* Patients presenting one or more of the following situations of malnutrition or nutritional risk: BMI <21 kg/m2 (or<23 kg/m2 in patients ≥ 65); unintentional weight loss >10% in the past 6 months; unintentional weight loss >5% in last moth; FFMI <15 kg/m2 (women) or <16 kg/m2 (men).
* Patients who signed informed consent.

Exclusion Criteria:

* Clinically unstable patients.
* Patients requiring other nutritional supplements or parenteral nutrition.
* Patients diagnosed with active pulmonary tuberculosis.
* Patients with acute respiratory failure.
* Patients with immunosuppression (including HIV, diabetes or neoplasms).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes in nutritional status | At hospital discharge or at 1th month and at 3 months
  Differences in weight, body mass index and fat free mass index evaluated by anthropometric measures.
Changes in pulmonary function | At 3rd month
  Differences in forced expiratory volume measured by spirometry.

SECONDARY OUTCOMES:
Respiratory Infections | At 1st, 2nd, 3rd month
  Differences measured by number of infections and hospital readmission rate.
Muscular Strength | At 3rd month.
  Differences measured by hand-grip strength.
Exercise Tolerance | At 3th month
  Differences measured by six minutes walk test.
Quality of Life of the participants | At hospital discharge or 1st month and 3rd month
  Differences measured by Saint George respiratory questionnaire.
Tolerability of the product | At 1st, 2nd and 3rd months
  Measured by gastrointestinal discomfort and product compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Antonio Camere Torrealva, Doctor, Principal Investigator — Clínica San Gabriel - Perú
Locations (1):
- Clínica San Gabriel, San Miguel, Lima region, Peru